CLINICAL TRIAL: NCT06571643
Title: Psoas Muscle Index (PMI) as a Predictor of Mobilisation and Postoperative Length of Stay After Minimally Invasive Cardiac Surgery
Brief Title: Psoas Muscle Index (PMI) as a Predictor of Outcomes After Minimally Invasive Cardiac Surgery
Acronym: PsoMICS
Status: Not yet recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: PsoMICS L2097
Record Dates: First submitted 2024-05-16; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Sarcopenia; Heart Valve Diseases
Keywords: Minimally invasive cardiac surgery; Psoas Muscle Index
MeSH Terms: conditions — Sarcopenia; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Lower Abdomen MRI — The patients will undergo a lower abdomen MRI to assess the size of the psoas muscle and derive the PMI

SUMMARY:
Sarcopenia or muscle loss and function is a component of the frailty syndrome. In this sense, frailty is becoming an important risk factor in predicting outcomes after major surgery and is defined as a geriatric syndrome of decreased reserve and resiliency to stressors that have been associated with adverse health outcomes in older adults. Despite its potentially relevant role in predicting postoperative recovery, frailty is rarely evaluated before surgery, and this is partially due to the low reliability of the most used frailty scores. Therefore, improvement in the frailty evaluation would be beneficial during the preoperative assessment of major surgeries. Sarcopenia, or the decline of skeletal muscle tissue with age, is one of the most important causes of functional decline and loss of independence in older adults and low muscle mass is a core component of frailty that has the advantage of being objectively quantifiable regardless of mobility, disability, or illness acuity. Psoas Muscle (PM) mass is an important parameter for evaluating muscle mass and has been previously correlated to frailty with a negative impact on the postoperative outcomes after major surgery and Psoas Muscle mass Index (PMI) is an easily available parameter for evaluating muscle mass and has already been demonstrated to be effective in predicting outcomes in different clinical settings. PMI has also been shown to be an effective predictor of outcomes in cardiac surgery although there are no studies specifically focusing on minimally invasive cardiac surgery. With this study, the investigators aim to investigate the relevance of PMI as a predictor of postoperative mobilisation, hospital length of stay and clinical recovery after major cardiac surgery conducted via a minimally invasive approach.

DETAILED DESCRIPTION:
This is a prospective, controlled, observational single-centre study of patients undergoing minimally invasive heart valve surgery at the department of minimally invasive cardiac surgery of the IRCCS Galeazzi Sant'Ambrogio Hospital, in Milan (Italy).

The primary endpoint is to evaluate the role of psoas muscle index (PMI) in predicting length of stay and early mobility after heart valve surgery via a minimally invasive approach.

25 consecutive participants patients undergoing minimally invasive cardiac surgery will be assessed with a lower abdomen MRI before the surgery to evaluate the diameter of the psoas muscle and therefore assess the Psoas Muscle Index (PMI). Frailty will be evaluated using the PRISMA-7 questionnaire.

PMI value will be correlated with the main outcomes via regression methods and adjusted for covariates.

The participants will be consented to the study before the cardiac surgery operation (indexed procedure). Surgeries will include aortic, mitral and tricuspid valve operations conducted either via a mini-thoracotomy or a mini-sternotomy approach and every patient will receive routine preoperative, operative and postoperative cardiac surgery care. In addition to standard cardiac surgery clinical variables, the investigators will collect data on:

* Total intubation hours
* Total Intensive Treatment Unit (ITU) length of stay
* Total postoperative length of hospital stay
* Time between end of surgery and first mobilisation (see below)

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (≥ 65 years old)
* Able to take consent
* Listed for minimally invasive cardiac surgery
* Elective and urgent procedures included
* Able to undergo MRI

Exclusion Criteria:

* Full median sternotomy approach
* Emergency procedures
* Unable to take consent
* Unable to undergo MRI

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Cardiac surgery patients undergoing heart valve surgery via a minimally invasive approach
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Intensive care unit (ITU) stay | perioperatively/periprocedurally
  Total number of hours spent in ITU after the primary (indexed) cardiac operation
Postoperative overall length of stay | perioperatively/periprocedurally
  Total number of days spent in hospital after the primary (indexed) cardiac operation
Mobilization time | perioperatively/periprocedurally
  Time to mobilization after the primary (indexed) cardiac operation defined as standing up or sitting down for at least 3 consecutive hours

SECONDARY OUTCOMES:
Postoperative mortality | perioperatively/periprocedurally
  In hospital mortality after the primary (indexed) cardiac operation
Long term mortality | at 1 year
  Mortality at the latest follow up after the primary (indexed) cardiac operation
Postoperative Complications | at 30 days
  Any surgical related postoperative complication related to the primary (indexed) cardiac operation

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy

REFERENCES:
- [Background] Benedek Z, Todor-Boer S, Kocsis L, Bauer O, Suciu N, Coros MF. Psoas Muscle Index Defined by Computer Tomography Predicts the Presence of Postoperative Complications in Colorectal Cancer Surgery. Medicina (Kaunas). 2021 May 11;57(5):472. doi: 10.3390/medicina57050472. PMID 34064607
- [Background] Bruno VD, Zakkar M. Psoas muscle index: a novel instrument in planning the treatment of severe aortic stenosis in frail patients. J Thorac Dis. 2018 Nov;10(Suppl 33):S4156-S4158. doi: 10.21037/jtd.2018.10.80. No abstract available. PMID 30631580
- [Background] Hawkins RB, Mehaffey JH, Charles EJ, Kern JA, Lim DS, Teman NR, Ailawadi G. Psoas Muscle Size Predicts Risk-Adjusted Outcomes After Surgical Aortic Valve Replacement. Ann Thorac Surg. 2018 Jul;106(1):39-45. doi: 10.1016/j.athoracsur.2018.02.010. Epub 2018 Mar 9. PMID 29530777
- [Background] Mamane S, Mullie L, Piazza N, Martucci G, Morais J, Vigano A, Levental M, Nelson K, Lange R, Afilalo J. Psoas Muscle Area and All-Cause Mortality After Transcatheter Aortic Valve Replacement: The Montreal-Munich Study. Can J Cardiol. 2016 Feb;32(2):177-82. doi: 10.1016/j.cjca.2015.12.002. Epub 2015 Dec 9. PMID 26821840
- [Background] Okamura H, Kimura N, Tanno K, Mieno M, Matsumoto H, Yamaguchi A, Adachi H. The impact of preoperative sarcopenia, defined based on psoas muscle area, on long-term outcomes of heart valve surgery. J Thorac Cardiovasc Surg. 2019 Mar;157(3):1071-1079.e3. doi: 10.1016/j.jtcvs.2018.06.098. Epub 2018 Jul 27. PMID 30139644
- [Background] Paknikar R, Friedman J, Cron D, Deeb GM, Chetcuti S, Grossman PM, Wang S, Englesbe M, Patel HJ. Psoas muscle size as a frailty measure for open and transcatheter aortic valve replacement. J Thorac Cardiovasc Surg. 2016 Mar;151(3):745-751. doi: 10.1016/j.jtcvs.2015.11.022. Epub 2015 Nov 21. PMID 26896357
- [Background] Raiche M, Hebert R, Dubois MF. PRISMA-7: a case-finding tool to identify older adults with moderate to severe disabilities. Arch Gerontol Geriatr. 2008 Jul-Aug;47(1):9-18. doi: 10.1016/j.archger.2007.06.004. Epub 2007 Aug 27. PMID 17723247
- [Background] Rodge GA, Goenka U, Jajodia S, Agarwal R, Afzalpurkar S, Roy A, Goenka MK. Psoas Muscle Index: A Simple and Reliable Method of Sarcopenia Assessment on Computed Tomography Scan in Chronic Liver Disease and its Impact on Mortality. J Clin Exp Hepatol. 2023 Mar-Apr;13(2):196-202. doi: 10.1016/j.jceh.2022.12.002. Epub 2022 Dec 9. PMID 36950487
- [Background] Walston JD. Sarcopenia in older adults. Curr Opin Rheumatol. 2012 Nov;24(6):623-7. doi: 10.1097/BOR.0b013e328358d59b. PMID 22955023
- [Background] Xu JY, Li C, Zhang H, Liu Y, Wei JM. Total Psoas Area Index is Valuable to Assess Sarcopenia, Sarcopenic Overweight/Obesity and Predict Outcomes in Patients Undergoing Open Pancreatoduodenectomy. Risk Manag Healthc Policy. 2020 Jul 9;13:761-770. doi: 10.2147/RMHP.S257677. eCollection 2020. PMID 32753989
- [Background] Wu XL, Shen J, Danzeng CD, Xu XS, Cao ZX, Jiang W. CT psoas calculations on the prognosis prediction of emergency laparotomy: a single-center, retrospective cohort study in eastern Asian population. World J Emerg Surg. 2022 Jun 3;17(1):31. doi: 10.1186/s13017-022-00435-x. PMID 35655215
- [Background] Yamashita M, Kamiya K, Matsunaga A, Kitamura T, Hamazaki N, Matsuzawa R, Nozaki K, Tanaka S, Nakamura T, Maekawa E, Masuda T, Ako J, Miyaji K. Prognostic Value of Psoas Muscle Area and Density in Patients Who Undergo Cardiovascular Surgery. Can J Cardiol. 2017 Dec;33(12):1652-1659. doi: 10.1016/j.cjca.2017.10.009. Epub 2017 Oct 16. PMID 29173605
- [Background] Zuckerman J, Ades M, Mullie L, Trnkus A, Morin JF, Langlois Y, Ma F, Levental M, Morais JA, Afilalo J. Psoas Muscle Area and Length of Stay in Older Adults Undergoing Cardiac Operations. Ann Thorac Surg. 2017 May;103(5):1498-1504. doi: 10.1016/j.athoracsur.2016.09.005. Epub 2016 Nov 15. PMID 27863730